CLINICAL TRIAL: NCT00932048
Title: Effect of Atorvastatin on Vascular Inflammation in Type 2 Diabetes: Analysis With 18F-Fluorodeoxyglucose Positron Emission Tomography
Brief Title: Effect of Atorvastatin on Vascular Inflammation in Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Kyung Mook Choi, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R0709211
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes; Atherosclerosis
Keywords: Diabetes Mellitus; Statins; PET
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Diabetes Mellitus | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10mg once daily for 12 weeks
  Arms: Atorvastatin

SUMMARY:
Type 2 diabetes mellitus significantly increases the risk for the development of atherosclerosis. Recently, atherosclerosis imaging with 18F-FDG PET (18F-Fluorodeoxyglucose Positron Emission Tomography) is useful for tracking inflammation within plaque and monitoring the response to drug therapy

The purpose of this study is to determine whether FDG-PET is capable of detecting atherosclerotic vascular inflammation and monitoring the early effects of statins in type 2 diabetic patients. The usefulness of FDG-PET in risk stratification is also investigated.

DETAILED DESCRIPTION:
The early detection of vulnerable plaques is clinically important for risk stratification and also to provide early treatment. Inflammation is important in the both pathogenesis and outcome of atherosclerosis. Plaques containing numerous inflammatory cells, particular macrophages, have a high risk of rupture. Diabetes is a major risk factor for the development of atherosclerosis. Lipid-lowering therapy with statins significantly decreases cardiovascular morbidity and mortality in primary and secondary prevention. Statin exert their benefits through the inhibition of de novo cholesterol synthesis, resulting in significant reductions in plasma low-density lipoprotein cholesterol (LDL-C) levels. It remains controversial whether LDL-C lowering is the only mechanism for the observed beneficial effects. Many LDL-C-independent pleiotropic effects have been postulated. Moreover, Lipid lowering therapy may affect atherosclerosis also through the inhibition of inflammatory marker. These evidences highlight the possibility of statins could be have great impact on plaque inflammation. 18FDG is a glucose analogue that is taken up by cells in proportion to their metabolic activity. Several papers have reported the potential roles of metabolic imaging in the assessment of inflammatory vascular diseases, especially in large vessels. If so, FDG-PET can monitor the direct effect of statins on vascular inflammation. Additionally, monitoring the vascular inflammation by FDG-PET may be useful for determining the risk stratification of atherosclerotic patients. The investigators hypothesize that statins-induced attenuation of vascular inflammation could be monitored clinically by use of FDG-PET approach, and providing information of early efficacy statins therapy caused by stabilization of vulnerable plaque without affecting the lumen size.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients who are aged 35 to 80 year-old

Exclusion Criteria:

* Insulin use
* Patients who receive any dyslipidaemia under medications (including statins) in recent one year
* Women of child-bearing potential are excluded (i.e. menopausal women or post-hysterectomy women are included in this study) due to radiation exposure in this study
* Active inflammatory diseases
* Vasculitis, symptomatic coronary artery disease, symptomatic cerebrovascular diseases
* Significant concomitant disease such as active infection, malignancy, hepatic or renal dysfunction at the time of enrollment (i.e. T-Bil > 3 mg/dl，ALT > 2.5 times the upper limit of normal range and Creatinine > 2 mg/dl in our hospital)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Vascular inflammation analyzed by PET: Define attenuation of plaque inflammation (plaque SUV or TBR) at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Change in LDL-cholesterol levels after active treatment | 12 weeks
Biomarkers: hs-CRP, adiponectin, MCP-1, PAI-1, TNF-α, IL-6 | 12 weeks
Change in carotid plaque thickness by ultrasound | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD. PhD, Principal Investigator — Korea University
Locations (1):
- Tae Nyun Kim, Seoul, South Korea